CLINICAL TRIAL: NCT06366477
Title: Effects of Vibration Stimulation Combined With Task-oriented Training on Hand Motor Function in Chronic Stroke: a Case Series Study
Brief Title: Effects of Vibration Stimulation Combined With Task-oriented Training on Hand Motor Function in Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B-ER-103-417
Record Dates: First submitted 2024-03-29; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-03

CONDITIONS: Rehabilitation; Stroke; Hand Grasp
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vibration stimulation combined with task-oriented training (Experimental)
  Interventions: Device: Vibration stimulation combined with task-oriented training

INTERVENTIONS:
Device: Vibration stimulation combined with task-oriented training — Participants with chronic stroke underwent 24 sessions of vibration stimulation combined with task-oriented training over 12 weeks, in addition to regular therapy.

SUMMARY:
There is a lack of effective therapies for hand and finger function recovery in people with chronic stroke. This study assessed the effects of combining vibration stimulation with task-oriented training on functional recovery, and treatment persistence. Participants with chronic stroke underwent 24 sessions of vibration stimulation combined with task-oriented training over 12 weeks, in addition to regular therapy. Functional recovery was assessed using the Fugl-Meyer assessment for motor function (FMA-wrist and hand), the Box and Blocks Test (BBT) for hand dexterity, and the Motor Activity Log (MAL) for daily functional activities. Minimal detectable change (MDC) and minimal important difference (MID) criteria were applied to interpret changes in assessment scores.

ELIGIBILITY:
Inclusion Criteria:

* Hemiparesis after stroke
* At least 6 months post-stroke
* Aged between 20 and 80 years
* Upper extremity Brunnstrom stage IV or V
* In stable medical condition
* No cognitive deficits (able to understand and follow the instructions)

Exclusion Criteria:

* Sensory impairment which may limit the participation in vibration stimulation treatment
* Other neurological or musculoskeletal impairments
* More than 2 by the Modified Ashworth Scale (0-5)
* Skin problems that prohibit participants from wearing the vibratory gloves
* Aphasia
* Apraxia
* Received other treatments which may influence motor or sensory abilities
* Participating in other studies in the past 6 months

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer assessment - wrist and hand | At baseline, 1 month after the start of the treatment, 2 months after the start of the treatment, 3 months after the start of the treatment, 1 month after the treatment ends and 3 months after the treatment ends.
  Fugl-Meyer assessment - wrist and hand is used to assess wrist and hand motor impairments in people with post stroke hemiplegia. Scoring is conducted through the direct assessment of the individual's performance, whereby the 12 items on the scale are scored according to their level of completion using a 3-point ordinal scale: 0 indicating inability to perform, 1 indicating partial performance, and 2 indicating full performance. The minimum score is 0. The total score is 24. The higher the score, the better the hand and wrist motor function.
Box and Blocks Test | At baseline, 1 month after the start of the treatment, 2 months after the start of the treatment, 3 months after the start of the treatment, 1 month after the treatment ends and 3 months after the treatment ends.
  Box and Blocks Test is a test of manual dexterity to assess hand function. The minimum score is 0. The total score is based on the number of blocks transferred from one box to the other in 60 seconds. Higher score is indicative of better hand dexterity.
Motor Activity Log | At baseline, 1 month after the start of the treatment, 2 months after the start of the treatment, 3 months after the start of the treatment, 1 month after the treatment ends and 3 months after the treatment ends.
  The Motor Activity Log is a structured interview intended to measure an individual's real life functional affected upper limb performance. The Motor Activity Log consists of two subtests: one pertaining to the amount of use (AOU) and the other pertaining to the quality of movement (QOM) of the affected upper limb. The Motor Activity Log employs an 11-point Likert scale, ranging from 0 to 5 with half-point increments, to evaluate the AOU and QOM subtests. The scores for AOU vary from 0, indicating never use the affected limb for this activity, to 5, indicating always use. Similarly, the scores for QOM range from 0, representing an inability to use the affected limb during the activity, to 5, indicating an ability to use the affected limb just as proficiently as before the stroke. Higher scores represent better performance.
Quantitative Electroencephalography Analysis: Delta Brain Symmetry Index | At baseline, 3 months after the start of the treatment and 3 months after the treatment ends.
  The Delta Brain Symmetry Index is a quantitative electroencephalography analysis used to assess hemispheric power lateralization and reflect improvements in hand motor functions. Delta Brain Symmetry Index ranges from 0 to 1, with higher indices indicating greater asymmetry and lower indices indicating more symmetry. Decreased Delta Brain Symmetry indicates a decrease in lateralization, potentially associated with brain reorganization that supports motor recovery.

IPD SHARING:
Plan to Share IPD: No
Quantitative Electroencephalography (QEEG): changes in hemispheric power lateralization. Functional recovery was assessed using the Fugl-Meyer assessment for motor function (FMA-wrist and hand), the Box and Blocks Test (BBT) for hand dexterity, and the Motor Activity Log (MAL) for daily functional activities.